CLINICAL TRIAL: NCT05093595
Title: Trans-nasal ETT Fixation
Brief Title: the Effect of Trans-nasal Fixation of Endotracheal Tubes for Prone Ventilation
Acronym: Trans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yue Yun, Attending Doctor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019
Record Dates: First submitted 2021-10-12; First posted 2021-10-26 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-10

CONDITIONS: Prone Craniotomy; Endotracheal Intubation Fixation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): The tracheal tube was routinely fixed with a teeth pad and adhesive tape (3M).
- Group B (Experimental): The tracheal tube was fixed by the trans-nasal Silicone Foley Catheter (SFC) and adhesive tape.
  Interventions: Device: SFC

INTERVENTIONS:
Device: SFC — The lubricated SFC passed nasally into the oropharynx under the visual guidance of visual laryngoscope to ensure that the cuff had passed through the posterior choanae and reached the oropharynx. The guide wire is removed and the balloon inflated with 5 ml normal saline. The catheter is then pulled slightly until the balloon is fixed and concealed by the soft palate . The ETT is anchored to the SFC with a cable tie .
  Arms: Group B

SUMMARY:
The aim of this randomized controlled trial is to evaluate the clinical effects of trans-nasal ETT fixation for prone ventilation.

ELIGIBILITY:
Inclusion criteria

* age 18-60 years old,
* ASA grade Ⅰ-Ⅱ,
* 18<BMI<24.

Exclusion criteria

* the intubation time was less than 5 hours,
* oral and facial skin damage,
* allergic to adhensive tapes,
* nasotracheal intubation,
* patients were edentulous.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
the distance of tube movement | The participants will be followed from intubation to extubation, an expected average of 6 hours.
  It is the difference between the preoperative depth of the supine tracheal tube and the postoperative depth of the prone tracheal tube.

CONTACTS AND LOCATIONS:
Locations (1):
- Yue Yun, Shenyang, Liaoning, China